CLINICAL TRIAL: NCT06568835
Title: Effect of Active Exercise on Nutritional and Inflammatory Status, Muscle Metabolism and Cardiovascular Events in Maintenance Haemodialysis Patients
Brief Title: The Effect of Active Exercise on Maintenance Haemodialysis Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunfeng Xia (Other)
Responsible Party: Sponsor-Investigator, Yunfeng Xia, Doctor, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: First ChongQing MU
Record Dates: First submitted 2024-07-31; First posted 2024-08-23 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Renal Dialysis
Keywords: Exercise; Inflammation; Nutrition; Muscular Atrophy
MeSH Terms: conditions — Motor Activity; Inflammation; Muscular Atrophy | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Active exercise group: patients were asked to choose walking (no less than 8000 steps per day) or low-intensity aerobic exercise such as jogging, swimming, Tai Chi, etc., according to their own conditions, for no less than 30 minutes each time, at least 3 times per week, and the intensity of the exercise was determined by the need to increase the frequency and depth of breathing during the exercise, and it was appropriate to feel slightly tired but not exhausted (RPE score 12-16).
  Exercise intensity should be at least 3 times a week, and the exercise intensity should be at a level that requires an increase in breathing rate and depth, allowing for dialogue and communication, slight sweating, and a feeling of being slightly tired but not exhausted (RPE score of 12 to 16).
  Control group: only receive conventional MHD treatment, no requirement for exercise.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): patients were asked to choose walking (no less than 8000 steps per day) or low-intensity aerobic exercise such as jogging, swimming, Tai Chi, etc., according to their own conditions, for no less than 30 minutes each time, at least 3 times per week, and the intensity of the exercise was determined by the need to increase the frequency and depth of breathing during the exercise, and it was appropriate to feel slightly tired but not exhausted (RPE score 12-16).
  Exercise intensity should be at least 3 times a week, and the exercise intensity should be at a level that requires an increase in breathing rate and depth, allowing for dialogue and communication, slight sweating, and a feeling of being slightly tired but not exhausted (RPE score of 12 to 16).
  Interventions: Behavioral: exercise
- Control group (No Intervention): only receive conventional MHD treatment, no requirement for exercise.

INTERVENTIONS:
Behavioral: exercise — such as walking, jogging, swimming, Tai Chi, etc. It needs to be at a certain frequency and intensity
  Arms: exercise group

SUMMARY:
The goal of this clinical trial is to discuss the effects of physical activity on nutrition, inflammation, muscle metabolism, and the occurrence of cardiovascular and cerebrovascular events in patients with maintenance haemodialysis. The main question it aims to answer is: can exercise improve nutritional and inflammatory status, enhance muscle strength, and reduce the incidence of cardiovascular and cerebrovascular events in patients with maintenance haemodialysis.

Researchers will compared active exercise group to conventional treatment group to see the impact of exercise on maintenance haemodialysis patients.

Participants will:

Choose low-intensity aerobic exercise workouts such as walking (no less than 8,000 steps per day) or jogging, swimming, Tai Chi, etc., according to their individual conditions, for no less than 30 minutes at a time, at least 3 times per week, and the intensity of the exercise should be based on an RPE score of 12 to 16.

DETAILED DESCRIPTION:
RPE: Rating of Perceived Exertion. RPE scores of 12 to 16 indicate the need for increased respiratory rate and depth during exercise, the ability to engage in conversational exchanges, light sweating, and a feeling of slight fatigue without reaching a state of exhaustion.

ELIGIBILITY:
Inclusion Criteria:

* MHD more than 3 months, 3 times per week, 3-4h each time;
* Urea clearance index (Kt/V) >1.2;
* Stable condition, no serious infection, tumour and cardiovascular disease;
* Willing to join the study and sign the informed consent form.

Exclusion Criteria:

* Combined with serious heart and lung disease: such as repeated heart failure, severe arrhythmia, unstable angina pectoris, severe pericardial effusion, severe heart valve disease, hypertrophic cardiomyopathy, aortic coarctation, severe emphysema, pulmonary heart disease, severe pulmonary hypertension (average pressure of the pulmonary artery > 55mmHg), etc.;
* Combined with chronic joints, muscles, or vascular disease can not be or is not suitable for regular exercise, such as cerebrovascular disease; combined chronic joint, muscle or vascular disease can not or are not suitable for regular exercise, such as cerebrovascular disease sequelae, serious lower limb joint damage, severe myopathy, deep vein thrombosis, etc.;
* unwilling to cooperate with the movement of people

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Mid-upper arm circumference of the non-internal fistula side（AC） | Baseline and half year, 1 year
  Measure the circumference of the non-internal fistula at the midpoint of the upper arm using a soft tape measure, in centimetres
triceps skin-fold thickness of the non-internal fistula side（TSF） | Baseline and half year, 1 year
  Measurement of the skinfold at the midpoint of the upper arm on the non-internal fistula side by using a skinfold thickness gauge, in centimetres
upper arm muscle circumference of the non-internal fistula side（AMC） | Baseline and half year, 1 year
  AMC（cm）= AC(cm) - 3.14 x TSF（cm）
calf circumference | Baseline and half year, 1 year
  Measure the calf circumference using a soft tape measure, in centimetres
grip strength | Baseline and half year, 1 year
  Using a grip strength meter, with the patient seated and gripping the handle firmly with the palm of the non-internal fistulae side, measure twice and record the maximum grip strength value
Incidence of cardiovascular and cerebrovascular events | 1 year
  Cardiovascular events include: heart failure episodes, sustained arrhythmias, myocardial infarction, and cerebrovascular events include: cerebral haemorrhage, cerebral infarction, transient ischaemic attack.

SECONDARY OUTCOMES:
prealbumin | Baseline and half year, 1 year
  laboratory measurement indicators:prealbumin(g/L)
albumin | Baseline and half year, 1 year
  laboratory measurement indicators:albumin(g/L)
haemoglobin | Baseline and half year, 1 year
  laboratory measurement indicators:haemoglobin(g/L)
blood lipids | Baseline and half year, 1 year
  laboratory measurement indicators:triglycerides, cholesterol, low-density lipoprotein, high-density lipoprotein
c-reactive protein | Baseline and half year, 1 year
  laboratory measurement indicators:c-reactive protein(mg/L)

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No